CLINICAL TRIAL: NCT03054558
Title: Predictive Value of Junctional Zone Thickness in Combination With Three Dimensional Power Doppler and Uterine Artery Vascular Indices in Patients With Recurrent Unexplained Pregnancy Loss; A New Diagnostic Tool.
Brief Title: JZ Thickness as a Predictor of Recurrent Unexplained First Trimesteric Pregnancy Loss.
Acronym: JZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: sherine Hosny Mohamed Gad Allah (Other)
Responsible Party: Sponsor-Investigator, sherine Hosny Mohamed Gad Allah, Assisstant professor of obs and gyne cairo uneveristy ,MD, Cairo University
Organization: Cairo University (Other)
Other Study IDs: C111
Record Dates: First submitted 2017-02-11; First posted 2017-02-15 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Patients With Recurrent Unexplained Pregnancy Loss
Keywords: Junctional zone; recurrent pregnancy loss; 3D power Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patients with recurrent unexplained pregnancy loss: Patients with history of two or more recurrent pregnancy loss (RPL) and no history of living babies who had performed all investigations for recurrent miscarriage (RM) including : laboratory investigation ,trans vaginal ultrasound (TVS) ,autoimmune work up and hystroscopy and all results were free
  Interventions: Other: Pelvic ultrasound both two dimensional and three dimentional
- Healthy fertile patients: Healthy fertile patients with no history of previous miscarriage and have at least one uncomplicated pregnancy with no pelvic pathology
  Interventions: Other: Pelvic ultrasound both two dimensional and three dimentional

INTERVENTIONS:
Other: Pelvic ultrasound both two dimensional and three dimentional

SUMMARY:
Patients with history of two or more recurrent pregnancy loss (RPL) and no history of living babies who had performed all investigations for recurrent miscarriage (RM) including : laboratory investigation ,trans vaginal ultrasound (TVS) ,autoimmune work up and hystroscopy and all results were free,will be scheduled for three dimensional trans-vaginal ultrasound (3D TVS) in the midluteal phase for measuring the impedance of uterine artery blood flow( by two dimensional Power Doppler TVS).Also by using 3D power Doppler the sub-endometrial blood flow will be assessed. In addition to the thickness of Junctional Zone (JZ) by using coronal view of 3 D TVS. To be compared with patients who had at least one full term living baby through normal vaginal delivery with no history of early pregnancy loss.

DETAILED DESCRIPTION:
Among patients attending the Recurrent pregnancy loss outpatient clinic of kasr Al Aini teaching hospital, Cairo University .Those meeting investigators inclusion criteria will be selected for the study. All patients had a history of two or more consecutive, first trimester miscarriages. Patients with two miscarriages will be included in the study since equal frequencies of abnormal test results have been demonstrated among patients with two miscarriages or more . Accordingly, the American College of Obstetrics and Gynecologists states that the evaluation of couples with two consecutive miscarriages should be initiated.

All women will undergo an extensive examination ,investigations (laboratory ,TVS and hystroscopy) in order to evaluate all known etiological factors for RPL.

Only Patients with free examination and normal investigations will be enrolled in our study.

Healthy fertile women who attended the outpatient clinic of obstetrics and gynecology in kasr Al Aini hospital ,Cairo university,for a routine scan will be recruited for the control group. Inclusion criteria required the absence of previous miscarriages and the presence of at least one previous uncomplicated pregnancy. Women with a history of pelvic disease or with abnormal findings during the ultrasound examination were excluded from the study.

The thickness and the morphology of the JZ will be evaluated on the uterine coronal view obtained by 3D TVS. Endometrial thickness with be measured and subendometrial blood flow ( vascularization index VI ,flow index FI and vascularization flow index VFI ) will be obtained by 3D power Doppler .

The sonographic evaluation will be performed in the midluteal phase of the cycle (18th to 22nd cycle day), to avoid possible hormonal influences, using an E8 (GE Healthcare, Zipf, Austria) ultrasound machine equipped with a multifrequency 3D volume endovaginal probe (2.8-10 MHz).

The examination included a 2D-TVS evaluation of the pelvic organs to exclude any abnormalities. Transvaginal Doppler flow measurement of the impendence to uterine artery blood flow was performed.

In order to evaluate the JZ the coronal view of the uterus will be obtained using 3D-TVS. Two to four static grey-scale volumes of the uterus will be obtained from the sagittal plane and from the transverse plane. The volume acquisition technique will be performed in a standardized fashion.

Recent studies indicate that the use of these criteria allow to an assessment of the JZ reproducible enough to be used in clinical practice. In particular: frequency, 6-9 MHz; magnification of the uterus up to half of the screen; sweep angle, 1208; sweep velocity will be adjusted from medium to maximum quality; 3D volume box exceeding the uterus by 1 cm on each side.

The coronal view reconstruction technique involved placing a straight or curved line (OmniView or rendering mode) along the endometrial stripe on the sagittal and transverse views. The multiplanar view was then manipulated until a satisfactory coronal image is obtained of the uterine external profile and the cavity, with bilateral visualization of the interstitial portion of the Fallopian tube. Volume contrast imaging (VCI) is applied (2- 4 mm slice thickness) with volume rendering (mixed light surface and gradient light). Following acquisition, ultrasound volumes will be stored for subsequent offline analysis. On the coronal view the JZ appears as a hypo-echoic zone around the endometrium. JZ measurements are therefore performed only on 3D multi-planar view using VCI. Disruption and infiltration of the hypo-echoic JZ by the hyper-echoic endometrial tissue are evaluated and the JZ thickness is measured as the distance from the basal endometrium to the internal layer of the outer myometrium. The minimum (JZmin), the maximum (JZmax) and the difference between the maximum and the minimum JZ (JZmax - JZmin) thickness are assessed. The JZmax and the JZmin are defined as the largest and smallest JZ thickness measured on a coronal or longitudinal section at any level of the uterus (fundus or anterior, posterior or lateral walls).

ELIGIBILITY:
Inclusion Criteria:

* Females with history of recurrent pregnancy loss
* for control group healthy females with history of at least one uncomplicated full pregnancy.

Exclusion Criteria:

* no history of endocrinal disorders
* no history of immunological diseases
* no history of pelvic pathology
* no history of uterine anomalies or cervical incompetence As a cause of recurrent pregnancy loss

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young females with history of two or more consecutive unexplained pregnancy loss who attend Kasr alainy out patient clinic seeking for fertility..
  Control group are healthy females of the same age group with no history of pregnancy loss and history of at least one full term healthy pregnancy who attends outpatient clinic for routine check up
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Thickness of junctional zone | immediatly measured by 3D TVS
  Measured in coronal view of 3DTVS

SECONDARY OUTCOMES:
Uterine artery Doppler Indices | immediatly measured by 2D power Doppler TVS
  measuring uterine artery pulsativity index (PI)
Subendometrial blood flow | immediatly measured by 3d power Doppler TVS
  Measuring flow index (FI) ,vascularization index(VI) and vascularization flow index(VFI)
Endometrial thickness | immediatly measured by 2D power Doppler TVS
  measuring endometrial thickness by 2d TVS (longitudinal view)

CONTACTS AND LOCATIONS:
Overall Officials: Sherine H Gad Allah, MD, Principal Investigator — kasr al aini teaching hospital
Locations (1):
- Kasr AlAini teaching hospital, Cairo, Egypt